CLINICAL TRIAL: NCT02080897
Title: Evaluating Quality of Life in Patients With Soft Tissue Sarcoma Presenting With Metastatic Lung Disease Using the ESAS-Sarcoma Modified Questionnaire
Brief Title: Evaluating Quality of Life in Patients With Soft Tissue Sarcoma Presenting With Metastatic Lung Disease
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00044852
Record Dates: First submitted 2014-03-05; First posted 2014-03-07 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Soft Tissue Sarcoma; Metastatic Lung Disease
Keywords: non-surgical; palliative surgery
MeSH Terms: conditions — Sarcoma; Lung Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Palliative Surgery Group: Patients who present to clinic with soft tissue sarcoma with metastatic lung disease who opt to proceed with palliative surgical treatment
- Non-surgical Group: Patients who present to clinic with soft tissue sarcoma with metastatic lung disease who opt not to pursue palliative surgery

SUMMARY:
The purpose of this study is to evaluate the role of palliative surgery in improving Quality of Life (QoL) and symptom control for patients who present with a Soft Tissue Sarcoma (STS) and metastatic lung disease. Responses to clinical Edmonton Symptom Assessment System - Sarcoma Modified ( ESAS-SM) questionnaire for patients who have undergone surgery for resection of the primary tumour will be compared to those that are unable to have surgery. Data collected from this questionnaire can highlight the benefits in patients' QoL who receive palliative surgical resection, and whether these benefits surmount those who are not treated with palliative surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with soft tissue sarcoma with at least one pulmonary metastasis
* Metastatic lung disease must have been present at time of initial presentation

Exclusion Criteria:

* All patients under 18 will be excluded
* Patients who have been previously undergone surgical resection of the primary tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with soft tissue sarcoma with metastatic lung disease
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2014-03; Primary Completion 2017-08-07 (Actual); Study Completion 2017-08-07 (Actual)

PRIMARY OUTCOMES:
Change in QoL score using patient-response questionnaire | questionnaire will be obtained at initial presentation and at up to 7 additional visits (6 weeks, 3 months, 6 months, 12 months, 24 months, 36 months and 60 months after initial presentation or treatment)
  The Edmonton Symptom Assessment System - Sarcoma Modified ( ESAS-SM) questionnaire will be completed at baseline, 6 weeks and 3, 6, 12, 24, 36 and 60 months post presentation/surgical intervention.

CONTACTS AND LOCATIONS:
Overall Officials: William Eward, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States